CLINICAL TRIAL: NCT03800225
Title: Treatment of Anterior Ligament Rupture With Internal Brace Repair - A Prospective Randomised Controlled Study Comparing Internal Brace Repair and a Patella Tendon Autograft Reconstruction.
Brief Title: Treatment of Anterior Ligament Rupture With Internal Brace Repair - A Prospective Randomised Controlled Study.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: A new scientific study shows that surgery with internal brace is worse than convensional surgery tecnic. This new knowledge stops this trial.
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Martin Lind, Professor, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Danish EC - 1-10-72-223-18.
Record Dates: First submitted 2019-01-09; First posted 2019-01-11 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Ligament; Laxity, Knee; Anterior Cruciate Ligament Injury
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Wound Healing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Repair (Experimental): Anterior cruciate ligament repair with internal brace after anterior ligament rupture.
  Interventions: Procedure: Repair
- Patella tendon graft (Active Comparator): The Patella tendon graft is harvested and used as a knew anterior cruciate ligament after rupture.
  Interventions: Procedure: Repair

INTERVENTIONS:
Procedure: Repair — Anterior ligament repair with internal brace.

SUMMARY:
The purpose of this study is to determine whether anterior cruciate ligament injury in patients wishing to return to sports activities may be treated with repair supplemented with internal brace compared with a standard operation using a patella tendon autograft.

ELIGIBILITY:
Inclusion Criteria:

* Anterior cruciate ligament rupture

Exclusion Criteria:

* Current malignant disease
* Rheumatoid arthritis
* Other knee ligament instability
* Obesity BMI >30
* Morbus Bechterew

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2019-09-04 (Actual); Study Completion 2019-09-04 (Actual)

PRIMARY OUTCOMES:
Knee Laxity | 12 Months
  KT-1000 arthrometer

SECONDARY OUTCOMES:
Patient reported outcome scores | 12 Months
  Koos (Knee injury and Osteoarthritis Outcome Score)
Patient reported outcome scores | 12 Months
  IKDC (International Knee Documentation Committee)
Pain measurement | 12 Months
  NRS-pain score (Numeric rating scale) (10 worst pain - 0 No pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Sports Trauma, Palle Juul-Jensens Boulevard 99, Aarhus N, Denmark